CLINICAL TRIAL: NCT05604508
Title: Testing Legally Feasible Options at Retail Point of Sale - Prices and Posters
Brief Title: Testing Legally Feasible Options Studies 2/3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, William Shadel, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA236608studies23; R01CA236608 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Commerce

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Status Quo (Active Comparator): This condition will allow for many posters with pricing information to be displayed.
  Interventions: Other: Many posters with prices
- Reduced Poster (Experimental): This condition will allow for a reduced number of posters with pricing information to be displayed.
  Interventions: Other: Fewer posters, no price restrictions
- No price (Experimental): This condition will allow for many posters with no pricing information to be displayed.
  Interventions: Other: Many posters, no prices

INTERVENTIONS:
Other: Many posters with prices — No poster number or price restrictions
  Arms: Status Quo
Other: Many posters, no prices — No poster number restrictions, but price restrictions
  Arms: No price
Other: Fewer posters, no price restrictions — Poster number restrictions, but no price restrictions
  Arms: Reduced Poster

SUMMARY:
The overall aim of this research is to experimentally evaluate different, legally-viable approaches to reducing the impact of the point-of-sale (POS) retail environment on adolescent tobacco use risk. This study will be investigating regulations for four classes of tobacco products (cigarettes, e-cigarettes, smokeless tobacco, little cigars/cigarillos). Study 2 and study 3 (out of 3 studies), occurring concurrently, will examine whether changing the number and content of posters on the outside doors at POS reduced adolescents' tobacco use risk.

DETAILED DESCRIPTION:
Tobacco advertising at retail point-of-sale (POS) includes promotional allowances that permit tobacco products to be advertised and sold at reduced cost to consumers (e.g., two-for-one specials); high visibility sale and therefore placement of hundreds of tobacco products on power walls; and the display of a large, diverse collection of poster advertisements on the exterior of the stores. Adolescents are at significant risk for having repeated exposures to this tobacco rich POS environment and such exposures contribute to increases in adolescent tobacco use. Although curbing the effect of the tobacco rich POS environment on adolescent tobacco use is a critical public health goal, some POS advertising regulations are unlikely to be viable in the United States because they impinge upon the tobacco industry's commercial free speech rights. For example, eliminating the tobacco power wall is probably not a viable option in the US as it has been successfully challenged in court by the tobacco industry. POS regulations that do not violate the industry's commercial free speech rights stand a better chance of being upheld by the courts. For example, eliminating tobacco product price promotions, reducing the availability of tobacco products by restricting the sale of flavored products, and restricting how much door/window space tobacco product posters can occupy at POS, all have been implemented as feasible and legally defensible regulatory options at POS. The evidence base supporting the efficacy of these initiatives is, however, almost non-existent - leaving them open to legal scrutiny. The overall aim of this research is to experimentally evaluate different, legally-viable approaches to reducing the impact of the POS retail environment on adolescent tobacco use risk. This research will be investigating the regulations for four classes of tobacco products (cigarettes, e-cigarettes, smokeless tobacco, little cigars/cigarillos): the extent to which eliminating tobacco product price promotions (Study 2), restricting how much door/window space tobacco posters can occupy at POS (Study 3), and eliminating the sale of flavored and/or mentholated tobacco products (Study 1) reduce adolescent tobacco-use risk. Each study will evaluate for possible gender and race (African-American vs Caucasian) differences. The studies will take place in the RAND StoreLab, a life-sized replica of a convenience store that was developed to experimentally evaluate how altering aspects of tobacco promotion at POS influences tobacco use. The present record is for Study 2 and Study 3.

ELIGIBILITY:
Inclusion Criteria:

ages 18-20, in college

-

Exclusion Criteria:

any medical or psychiatric condition which would make compliance with the study protocol difficult (based on parent report).

Previous participation in a previous StoreLab study

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 445 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RAND Corporation, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Status Quo | Reduced Poster | No Price
Started | 150 | 147 | 148
Completed | 150 | 147 | 148
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Status Quo | Reduced Poster | No Price | Total
Number analyzed (Participants) | 150 | 147 | 148 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some participants opted to not complete some information, hence the different n.
  years
    number analyzed (Participants) | 149 | 146 | 148 | 443
    (all) | 19.10 (0.77) | 19.16 (0.81) | 19.16 (0.78) | 19.14 (0.79)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Some participants opted to not enter demographic data.
  Participants
    Gender identity: number analyzed (Participants) | 149 | 146 | 148 | 443
    Gender identity: Male | 31 | 38 | 33 | 102
    Gender identity: Female | 102 | 98 | 106 | 306
    Gender identity: Other than male or female | 16 | 10 | 9 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some participants elected to not enter some demographic data.
  Participants
    number analyzed (Participants) | 149 | 145 | 147 | 441
    Hispanic or Latino | 12 | 18 | 11 | 41
    Not Hispanic or Latino | 137 | 127 | 136 | 400
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Some participants opted not to provide demographic information
  Participants
    number analyzed (Participants) | 148 | 146 | 148 | 442
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Asian | 51 | 55 | 51 | 157
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 15 | 17 | 8 | 40
    White | 72 | 66 | 75 | 213
    More than one race | 8 | 7 | 10 | 25
    Unknown or Not Reported | 2 | 0 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 150 | 147 | 148 | 445

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Cigarette Smoking Risk After Shopping in the StoreLab
Description: Respondents answer the following items: "Do you think you will try a cigarette anytime soon?", "Do you think you will try a cigarette anytime in the next year?"; and "If one of your best friends offered you a cigarette, would you smoke it?". Responses are made on a 1 (Definitely not) to 10 (Definitely yes) scale and summed to produce a total smoking risk scale score (range from 3 - 30). Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk). Outcome is proportion at risk of cigarette smoking (number of participants at risk over number of participants within condition).
Time Frame: There is one visit in this research: This variable is assessed at that visit, within 5 minutes of the experimental manipulation
Population: Some participants were missing data, which accounts for differences in the n.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Reduced Poster | No Price
Number analyzed (Participants) | 142 | 145 | 146
proportion of participants | .59 [.45 to .73] | .52 [.38 to .65] | .39 [.28 to .51]
Statistical Analysis 1: Comparison: Status Quo vs Reduced Poster; Test type: Other; Odds Ratio (OR) = 0.735, 95% CI 2-sided [0.347 to 1.553] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, and baseline cigarette use intentions
Statistical Analysis 2: Comparison: Status Quo vs No Price; Test type: Other; Odds Ratio (OR) = 0.471, 95% CI 2-sided [0.234 to 0.947] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, and baseline cigarette use intentions

2. Primary Outcome: Self-reported Vaping/ENDS Risk of Use
Description: Respondents answer the following items: "Do you think you will try a vaping product anytime soon?", "Do you think you will try a vaping product anytime in the next year?"; and "If one of your best friends offered you a vaping product, would you use it?". Responses are made on a 1 (Definitely not) to 10 (Definitely yes) scale and summed to produce a total vaping risk scale score (range from 3 - 30). Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk). Outcome is proportion at risk of vaping (number of participants at risk over number of participants within condition).
Time Frame: There is one visit in this research: This variable is assessed at that visit, within 5 minutes after experimental manipulation
Population: Some participants opted to not answer some items, hence the differing n.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Reduced Poster | No Price
Number analyzed (Participants) | 142 | 145 | 144
proportion of participants | 0.55 [0.40 to 0.69] | 0.68 [0.45 to 0.70] | 0.52 [0.37 to 0.67]
Statistical Analysis 1: Comparison: Status Quo vs Reduced Poster; Test type: Other; Odds Ratio (OR) = 1.503, 95% CI 2-sided [0.727 to 3.107] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, baseline vaping intentions
Statistical Analysis 2: Comparison: Status Quo vs No Price; Test type: Other; Odds Ratio (OR) = 0.878, 95% CI 2-sided [0.398 to 1.938] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, baseline vaping intentions

3. Primary Outcome: Self-reported Smokeless Tobacco Use Risk
Description: Respondents answer the following items: "Do you think you will use smokeless tobacco anytime soon?", "Do you think you will try smokeless tobacco anytime in the next year?"; and "If one of your best friends offered you smokeless tobacco, would you use it?". Responses are made on a 1 (Definitely not) to 4 (Definitely yes) scale and summed to produce a total smokeless tobacco risk scale score (range from 3 - 30). Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk). Outcome is proportion at risk of smokeless tobacco use (number of participants at risk over number of participants within condition).
Time Frame: as for outcome 1
Population: Some participants opted to not respond to some items, hence the different n.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Reduced Poster | No Price
Number analyzed (Participants) | 142 | 144 | 144
proportion of participants | 0.41 [0.28 to 0.54] | 0.30 [0.20 to 0.42] | 0.23 [0.14 to 0.34]
Statistical Analysis 1: Comparison: Status Quo vs Reduced Poster; Test type: Other; Odds Ratio (OR) = 0.619, 95% CI 2-sided [0.295 to 1.301] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, and baseline smokeless use intentions
Statistical Analysis 2: Comparison: Status Quo vs No Price; Test type: Other; Odds Ratio (OR) = 0.489, 95% CI 2-sided [0.237 to 1.006] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco, baseline smokeless use intentions

4. Primary Outcome: Self-reported Cigarillo/Little Cigar *LCC) Use Risk
Description: Respondents answer the following items: "Do you think you will try a cigarillo/little cigar anytime soon?", "Do you think you will try a cigarillo anytime in the next year?"; and "If one of your best friends offered you a cigarillo, would you smoke it?". Responses are made on a 1 (Definitely not) to 4 (Definitely yes) scale and summed to produce a total cigarillo risk scale score (range from 3 - 30). Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk). Outcome is proportion at risk of LCC use (number of participants at risk over number of participants within condition).
Time Frame: as for outcome 1
Population: Some participants opted to not complete some items, hence the different n.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Reduced Poster | No Price
Number analyzed (Participants) | 140 | 145 | 143
proportion of participants | 0.36 [0.24 to 0.49] | 0.41 [0.29 to 0.54] | 0.44 [0.31 to 0.58]
Statistical Analysis 1: Comparison: Status Quo vs Reduced Poster; Test type: Other; Odds Ratio (OR) = 1.428, 95% CI 2-sided [0.720 to 2.832] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, baseline LCC use intentions
Statistical Analysis 2: Comparison: Status Quo vs No Price; Test type: Other; Odds Ratio (OR) = 1.420, 95% CI 2-sided [0.681 to 2.960] — Adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, baseline LCC use intentions

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Status Quo | Reduced Poster | No Price
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/147 | 0/148
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/147 | 0/148
Other Adverse Events (participants affected / at risk) | 0/150 | 0/147 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT05604508/Prot_SAP_000.pdf